CLINICAL TRIAL: NCT01758133
Title: Influence of Medical Clown Activity on Milk Production of Mothers of Premature Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 006612-HYMC
Record Dates: First submitted 2012-12-24; First posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-12

CONDITIONS: Breast Milk

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Mothers exposed to medical clowns: Mothers of premature infants who have been exposed to medical clown activities
  Interventions: Behavioral: Exposure to medical clown activities
- Mothers not exposed to medical clown activity

INTERVENTIONS:
Behavioral: Exposure to medical clown activities
  Groups: Mothers exposed to medical clowns

SUMMARY:
The aim of this study is to determine whether medical clown activity enables relaxation of mothers of premature infants, and as a result increases their breast milk production.

ELIGIBILITY:
Inclusion Criteria:

* Nursing mothers of infants born less than 34th week

Exclusion Criteria:

* Sick mothers
* Take medication forbidden during nursing

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Mothers of premature infants
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Amount of breast milk produced | One week
  Mothers who have either been exposed or not exposed to medical clown activities will pump their breast milk. The milk will be measured and the two groups production will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel